CLINICAL TRIAL: NCT06795412
Title: A Phase 1/2, Open-label, Global, Multicenter, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of PYX-201 in Combination With Pembrolizumab in Participants With Advanced Solid Tumors
Brief Title: Study of PYX-201 in Combination With Pembrolizumab in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pyxis Oncology, Inc (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PYX-201-102; KEYNOTE-G17 (Other: Merck Sharp & Dohme LLC); MK-3475-G17 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumours
Keywords: Advanced Solid Tumours; PYX-201; Pembrolizumab
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive escalating doses of PYX-201 to evaluate the safety, tolerability, and preliminary efficacy of PYX-201 in combination with pembrolizumab.
  Interventions: Drug: PYX-201; Drug: pembrolizumab
- Part 2: Dose Expansion (Experimental): Part 2 dose-expansion cohorts will be opened based on emerging data to further inform the safety, tolerability, and preliminary efficacy determinations as defined.
  Interventions: Drug: PYX-201; Drug: pembrolizumab

INTERVENTIONS:
Drug: PYX-201 — Intravenous (IV) infusion.
Drug: pembrolizumab — IV infusion.
  Other Names: KEYTRUDA®

SUMMARY:
The primary objective of this study is to determine the recommended Phase 2 doses (RP2D(s)) and maximum tolerated dose (MTD) of PYX-201 in combination with pembrolizumab for participants with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed advanced solid tumors, including first-line (1L) head and neck squamous cell carcinoma (HNSCC), advanced or metastatic triple negative breast cancer (TNBC), hormone receptor positive (HR+) and human epidermal growth factor receptor 2 negative breast cancer (HER2- BC), gastric cancer (GC), cervical cancer, and second-line and higher (2L+) HNSCC.
2. Male or non-pregnant, non-lactating female participants age ≥18 years.
3. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1.
4. Participant must have at least 1 measurable lesion per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 criteria.
5. Life expectancy of >3 months, in the opinion of the Investigator.
6. Adequate hematologic function.
7. Adequate hepatic function.
8. Adequate renal function.
9. Adequate coagulation profile.
10. Clinical sites must conduct fresh tumor biopsy or provide participant's archived tumor tissue sample.

Exclusion Criteria

1. Known additional malignancy that is progressing or has required active treatment within the past 2 years.
2. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
3. Significant cardiovascular disease within 6 months prior to start of study drug.
4. Evidence of an active systemic bacterial, fungal, or viral infection requiring treatment at the start of study drug.
5. Known active hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS).
6. Failure to recover to Baseline severity or National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0 Grade ≤1 from acute non-hematologic toxicity due to previous therapy, prior to Screening.
7. Participants with active neuropathy of any grade per CTCAE v5.0 at Screening.
8. History of uncontrolled diabetes mellitus.
9. Participants with immunodeficiency or active autoimmune disease that is contraindicated for pembrolizumab.
10. Participants with a history of (noninfectious) pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD.
11. Prior solid organ or bone marrow progenitor cell transplantation.
12. Prior high-dose chemotherapy requiring stem cell rescue.
13. Previously received treatment with a programmed death-1 (PD-1)/L1 inhibitor any prior treatment with an agent directed to another stimulatory or co inhibitory T-cell receptor.
14. Severe hypersensitivity (Grade ≥3) to pembrolizumab and/or any of its excipients and/or PYX-201 and/or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2027-12-06 (Estimated); Study Completion 2027-12-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience a Dose-Limiting Toxicity (DLT) | Day 1 to Day 21
Number of Participants who Experience an Adverse Event (AE) | Up to approximately 2 years
Number of Participants who Experience Clinically Significant Changes in Clinical Laboratory Parameters | Up to approximately 2 years
Number of Participants who Experience Clinically Significant Changes in Vital Signs | Up to approximately 2 years
Number of Participants who Experience Clinically Significant Changes in electrocardiogram (ECG) Parameters | Up to approximately 2 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Day 1 up to approximately 2 years
Duration of Response (DOR) | Day 1 up to approximately 2 years
Disease Control Rate (DCR) | Day 1 up to approximately 2 years
Time to Response | Day 1 up to approximately 2 years
Clinical Benefit Rate (CBR) | Day 1 up to approximately 2 years
Maximum Observed Concentration (Cmax) of PYX-201 | Day 1 up to approximately 2 years
Time to Maximum Concentration (Tmax) of PYX-201 | Day 1 up to approximately 2 years
Clearance (CL) of PYX-201 | Day 1 up to approximately 2 years
Area Under the Concentration-time Curve from Time 0 to the Last Quantifiable Concentration (AUC0-t) of PYX-201 | Day 1 up to approximately 2 years
Area Under the Concentration-time Curve Over the Dosing Interval (AUCtau) of PYX-201 | Day 1 up to approximately 2 years
Area Under the Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC0-inf) of PYX-201 | Day 1 up to approximately 2 years
Half-Life (t½) for Antibody-drug Conjugate (ADC) | Day 1 up to approximately 2 years
Half-Life (t½) for Total Antibody (tAb) | Day 1 up to approximately 2 years
Half-Life (t½) for Free Payload | Day 1 up to approximately 2 years
Incidence of Anti-PYX-201 Antibodies | Day 1 up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California San Diego, San Diego, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Texas - M.D. Anderson Cancer Center, Houston, Texas
  - NEXT Oncology Houston, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No